CLINICAL TRIAL: NCT06342817
Title: Effects of a Meditation Program on the Sleep Quality of Medicine Course Students
Brief Title: Effects of Meditation on Sleep Quality of Medical Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal da Fronteira Sul (Other)
Responsible Party: Principal Investigator, Tiago Teixeira Simon, Tiago Teixeira Simon, Universidade Federal da Fronteira Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UFFS
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Sleep Disorder
Keywords: sleep disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Those students interested in participating in the study will leave their contact details (telephone and email) to the research coordinator, to whom it will be sent an online questionnaire containing the inclusion and exclusion criteria, and the free consent form through the Google forms platform. Collection instruments will only be made available after fulfilling the inclusion criteria and absence of exclusion criteria and agreement with the consent form. Responders will be randomly randomized 1:1 and subsequently communicated whether they will participate in the intervention group or the control group.
Masking Description: Responders will be randomly randomized 1:1 and subsequently communicated whether they will participate in the intervention group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will attend 8 weekly online meetings lasting approximately 60 minutes each (generally structured in an initial 10 minutes for questions about the practices, 15-20 minutes of exposition on the central theme of the meeting, 5-10 minutes for class practice, 10-15 minutes for post-practice inquiry, 5 minutes for explanation of the week's informal practice and audios for daily practice). Audio in mp3 of the practice carried out at each meeting will be provided to maintain daily individual practice during the week. An online questionnaire related to weekly practices will also be left at the beginning of each meeting.
  Interventions: Behavioral: online mindfulness based meditation program
- control group (No Intervention): In the control group there will be no intervention. Participants will only participate in the initial meeting explaining the study design and their role in it, inviting them to complete the questionnaires at the same time as the intervention group. They will commit to not receiving any intervention and will be asked not to participate in any meditation or mindfulness sessions during the period of application of the POMBM to the intervention group (8 weeks). After the end of this period, it will be offered the possibility to take the POMBM as they wish.

INTERVENTIONS:
Behavioral: online mindfulness based meditation program — Participants in the intervention group will attend 8 weekly online meetings lasting approximately 60 minutes each (generally structured in an initial 10 minutes for questions about the practices, 15-20 minutes of exposition on the central theme of the meeting, 5-10 minutes for class practice, 10-15 minutes for post-practice inquiry, 5 minutes for explanation of the week's informal practice and audios for daily practice). Audio in mp3 of the practice carried out at each meeting will be provided to maintain daily individual practice during the week. An online questionnaire related to weekly practices will also be left at the beginning of each meeting.
  Arms: Intervention

SUMMARY:
The objective of the study is to evaluate the effect of an 8-week online mindfulness-based meditation program on quality sleep status of undergraduate students medicine in the city of Passo Fundo/RS and Chapecó/SC In addition to sleep quality, secondary outcomes such as mindfulness, symptoms of depression, stress, anxiety and burnout will also be assessed

DETAILED DESCRIPTION:
A controlled, single-center, randomized parallel group clinical trial will be developed to evaluate the effectiveness of an online mindfulness-based meditation program (POMBM) on the quality of sleep of medical students. The trial expects to involve 136 participants who will be randomized 1:1 into the intervention group or a waiting group (which will be called the control group), with 68 expected participants each. All trial procedures will take place online via Google meet and will consist of an invitation and presentation of the study, followed by an initial screening visit for those interested, and an intervention period of 8 weeks. The POMBM will be administered weekly online during the intervention period, with each session lasting 45 to 60 minutes. The control group will not perform any activities during the intervention period. Participants in both groups will be evaluated at the initial visit (T0), in the fifth week (T1), immediately after the end of the intervention period (T2) and in a 2-month follow-up after the end of the program (T3) using the following instruments : PSQI (Pittsburgh Quality Sleep Index), ESE (Epworth Sleepiness Scale), MAAS (Mindful Attention Awareness Scale), DASS-21 (Depression, Anxiety and Stress Scale), and CBI-S (Copenhagen Burnout Inventory Student Version)

ELIGIBILITY:
Inclusion Criteria:

* Interest in participating in the study; over 18 years old; both genders; being duly registered in the Medicine course at Passo Fundo or Chapecó's faculties, from the 1st to 12th phase of the course

Exclusion Criteria:

* Have participated in another course or workshop on meditation in the last 4 weeks in addition to the invitation to study; being an active practitioner of meditation, yoga, tai-chi, qui-gong (at least 6 months before the start of the study); previous medical diagnosis of cognitive, language or communication deficits; alcohol dependence and other chemical substances; previous medical diagnosis of a disorder with risk of suicide or attempt of previous suicide; previous medical diagnosis of post-traumatic stress disorder; previous medical diagnosis of depressive disorder currently untreated; previous medical diagnosis of schizophrenia or delusional/hallucinatory disorders; previous medical diagnosis of social anxiety (difficulty being in a classroom)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the quality of sleep of medical students on weeks 5, 9 and 17 by the PSQI and ESE | week 0, week 5, week 9 and week 17
  - PSQI (Pittsburgh Quality Sleep Index) - instrument consisting of 19 self-report questions categorized into seven components, graduated in scores from zero (no difficulty) to three (severe difficulty). The components of the PSQI are: C1 subjective sleep quality, C2 sleep latency, C3 sleep duration, C4 habitual sleep efficiency, C5 sleep changes, C6 use of sleeping medications C7 daytime sleep dysfunction. The sum of the values attributed to the seven components varies from zero to twenty-one in the total questionnaire score, indicating that the higher the number, the worse the sleep quality. A total score greater than five indicates that the individual is experiencing major dysfunction in at least two components, or moderate dysfunction in at least three components. ESE (Epworth Sleepiness Scale). This is a self-administered questionnaire that assesses the probability of falling asleep in eight situations involving daily activities, some of which are known to be highly soporific. The

SECONDARY OUTCOMES:
Change in the awareness of medical students on weeks 5, 9 and 17 by the MAAS | week 0, week 5, week 9 and week 17
  MAAS (Mindful Attention Awareness Scale). It is a 15-item unidimensional measure of mindfulness. Each item is rated on a Likert scale between 1 (almost always) and 6 (almost never) in relation to the interviewee's daily experience. Higher scores reflect higher levels of dispositional mindfulness
Change in the depression, anxiety and stress symptoms of medical students on weeks 5, 9 and 17 by the DASS-21 | week 0, week 5, week 9 and week 17
  DASS-21 (Depression, Anxiety and Stress Scale) This is a questionnaire with 21 questions, which measure the intensity of behaviors and sensations experienced in the last seven days. It has the ability to simultaneously measure and distinguish depression, anxiety and stress. Each question is rated on a four-point Likert scale of frequency or severity of participants' experiences during the past week with the intention of emphasizing emotional states over these traits.
Change in the burnout symptoms of medical students on weeks 5, 9 and 17 by CBI-S | week 0, week 5, week 9 and week 17
  CBI-S (Copenhagen Burnout Inventory - Student version) is a 19-item self-report measure of burnout. To adapt the instrument to the students' context, when adapting the original format, the instrument was composed of the following dimensions: Personal Burnout (PB), Study-Related Burnout (SRB), Colleague-Related Burnout (CRB) and Student-Related Burnout. Teachers (TRB), the questions relating to the third dimension were duplicated, increasing the questionnaire to 25 questions. Five response options are used, in two domains: one for intensity and another for frequency

CONTACTS AND LOCATIONS:
Overall Officials: Tiago T Simon, Principal Investigator — Universidade Federal da Fronteira Sul
Locations (1):
- Universidade Federal Da Fronteira Sul, Passo Fundo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
There´s no plan of IPD sharing

REFERENCES:
- [Background] Azad MC, Fraser K, Rumana N, Abdullah AF, Shahana N, Hanly PJ, Turin TC. Sleep disturbances among medical students: a global perspective. J Clin Sleep Med. 2015 Jan 15;11(1):69-74. doi: 10.5664/jcsm.4370. PMID 25515274
- [Background] BARROS, V. V. DE et al. Validity evidence of the brazilian version of the Mindful Attention Awareness Scale (MAAS). Psicologia: Reflexão e Crítica, v. 28, n. 1, p. 87-95, mar. 2015.
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Pedro VD, Menna Barreto SS, Johns MW. Portuguese-language version of the Epworth sleepiness scale: validation for use in Brazil. J Bras Pneumol. 2009 Sep;35(9):877-83. doi: 10.1590/s1806-37132009000900009. English, Portuguese. PMID 19820814
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008. PMID 18283207
- [Background] CAMPOS, J. A. D. B.; CARLOTTO, M. S.; MARÔCO, J. Copenhagen Burnout Inventory - student version: adaptation and transcultural validation for Portugal and Brazil. Psicologia: Reflexão e Crítica, v. 26, n. 1, p. 87-97, 2013.
- [Background] Dawson AF, Brown WW, Anderson J, Datta B, Donald JN, Hong K, Allan S, Mole TB, Jones PB, Galante J. Mindfulness-Based Interventions for University Students: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Appl Psychol Health Well Being. 2020 Jul;12(2):384-410. doi: 10.1111/aphw.12188. Epub 2019 Nov 19. PMID 31743957
- [Background] Jiang A, Rosario M, Stahl S, Gill JM, Rusch HL. The Effect of Virtual Mindfulness-Based Interventions on Sleep Quality: A Systematic Review of Randomized Controlled Trials. Curr Psychiatry Rep. 2021 Jul 23;23(9):62. doi: 10.1007/s11920-021-01272-6. PMID 34297230
- [Background] Ong JC, Moore C. What do we really know about mindfulness and sleep health? Curr Opin Psychol. 2020 Aug;34:18-22. doi: 10.1016/j.copsyc.2019.08.020. Epub 2019 Aug 24. PMID 31539830
- [Background] Rusch HL, Rosario M, Levison LM, Olivera A, Livingston WS, Wu T, Gill JM. The effect of mindfulness meditation on sleep quality: a systematic review and meta-analysis of randomized controlled trials. Ann N Y Acad Sci. 2019 Jun;1445(1):5-16. doi: 10.1111/nyas.13996. Epub 2018 Dec 21. PMID 30575050
- [Background] Vignola RC, Tucci AM. Adaptation and validation of the depression, anxiety and stress scale (DASS) to Brazilian Portuguese. J Affect Disord. 2014 Feb;155:104-9. doi: 10.1016/j.jad.2013.10.031. Epub 2013 Oct 28. PMID 24238871
- Available data/document: Study Protocol — https://drive.google.com/file/d/1YWyRsHac1y9eqsmQXVHCsmYArWwAdMoq/view?usp=sharing
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1TfBgnmUMvF4tFJu-a1lGXlcawu0k5YeJ/view?usp=sharing